CLINICAL TRIAL: NCT02763683
Title: Investigations of Dementia in Parkinson Disease
Acronym: PIB
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201512032; R01NS075321 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Parkinsons
Keywords: Parkinsons Disease; PET Imaging; PIB; VAT; Dementia
MeSH Terms: conditions — Parkinson Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinsons Disease: Individuals with Parkinsons Disease
  Interventions: Radiation: PiB and VAT
- Healthy Controls: Individuals without Parkinsons Disease
  Interventions: Radiation: PiB and VAT

INTERVENTIONS:
Radiation: PiB and VAT — There is no intervention for this study. The PiB and VAT are used during the PET procedures to help to identify any excessive abnormal proteins in the brain.

SUMMARY:
The purpose of this study is to use a brain imaging method called Pittsburgh B (PIB) Positron Emission Tomography (PET) and Vesicular Cholinergic Transport (VAT) PET to determine dementia subtypes in patients with Parkinson disease (PD). The ultimate goal of this project is to be able to identify individuals with PD who are at risk of developing dementia, and to distinguish the underlying cause of dementia.

DETAILED DESCRIPTION:
The purpose of this study is to use a brain imaging method called PIB PET and VAT PET to determine dementia subtypes in patients with Parkinson disease (PD). The ultimate goal of this project is to be able to identify individuals with PD who are at risk of developing dementia, and to distinguish the underlying cause of dementia. The investigators will be including both PD and normal subjects in this study. This a long term study and we are considering including a total of 320 participants in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* PD patients must exhibit three of the following cardinal signs: rest tremor, rigidity, bradykinesia, or postural instability; or two of these features with one of the first three displaying asymmetry.

Exclusion Criteria:

* history of head trauma, major neurological or psychiatric diseases other than Parkinson disease and dementia, e.g. stroke, multiple sclerosis, depression or schizophrenia.
* severe systemic diseases.
* inability to lie still for 90 minutes.
* metallic implants, pacemakers, or any other contraindication to MRI.
* refusal to consent to brain donation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with and without Parkinson disease will be recruited from the Movement Disorders Center at Washington University, the St. Louis metro area, and throughout the midwest region.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2016-06; Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Investigations of Dementia in Parkinsons Disease | 2030
  The investigators will perform memory/thinking testing, Lumbar puncture (LP), Magnetic Resonance Imaging (MRI) and (PET) scans to help to determine the cause(s) of memory and thinking in Parkinson Disease.
  The memory and thinking testing by phone on average at 1.5 years through study completion and then in person on average at 3 years through study completion, this will help monitor if there is any decline in memory and thinking.
  The Lumbar Puncture is done on willing participants on average at 3 years through study completion to assess for any abnormal proteins and correlate these with any changes in memory and thinking.
  The MRI is done on average at 3 years through study completion for any abnormal signs or changes in regards to dementia at 3 years.
  The (PiB) & (VAT) PET scans will be performed on average at 3 years through study completion, which will be analyzed to assess for changes in regards to abnormal proteins and signs of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Perlmutter, MD, Principal Investigator — Washington University School of Medicine; MD, Principal Investigator
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data that has been published will be shared upon request.
Supporting Information: ICF
Time Frame: after publication of the results
Access Criteria: request from a legitimate investigator with a proposal sent to and approved by Joel S Perlmutter at Washington University.